CLINICAL TRIAL: NCT02291627
Title: Comparison of the Macintosh, Coopdech and AirTraq Laryngoscopes Using a Rigid Neck Collar in Pediatric Patients With Simulated Difficult Laryngoscopy.
Brief Title: Pediatric Intubation With Difficult Airway
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/15
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Trauma; Intubation, Endotracheal
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intubation with immobilized cervical spine (Experimental): endotracheal intubation with immobilized cervical spine
  Interventions: Device: MAC; Device: Coopdech; Device: AirTraq

INTERVENTIONS:
Device: MAC — direct laryngoscopy
  Other Names: Macintosh Laryngoscope
Device: Coopdech — Video laryngoscopy
  Other Names: Coopdech Video Lartyngoscope Portable VLP-100
Device: AirTraq — optical laryngoscopy

SUMMARY:
The aim of this study was to compare time, success rates of different video laryngoscopes for the emergency intubation with an immobilized cervical spine in a standardized pediatric manikin model.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study
* minimum 1 year of work experience in emergency medicine
* experienced emergency medical personnel (physicians, nurses, paramedics)

Exclusion Criteria:

* Not meet the above criteria
* Wrist or Low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Success of intubation | 1 day
  effectiveness of first, second and third intubation attempts and overall effectiveness of intubation by participants

SECONDARY OUTCOMES:
Intubation time | 1 day
  time in seconds required for a successful intubation attempt
Cormack-Lehane grading | 1 day
  self-reported percentage the vocal cord visualization using the Cormack-Lehane grading (grade 1-4)

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland